CLINICAL TRIAL: NCT01049607
Title: Clamp-Crushing vs. Stapler Hepatectomy for Transection of the Parenchyma in Elective Hepatic Resection: CRUNSH - A Randomized Controlled Trial
Brief Title: Stapler Hepatectomy for Elective Liver Resection
Acronym: CRUNSH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nuh Rahbari (Other)
Responsible Party: Sponsor-Investigator, Nuh Rahbari, M.D. Resident, Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NNR-03
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Hepatic Resection
Keywords: Patients undergoing hepatic resection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clamp-Crush technique (Active Comparator)
  Interventions: Procedure: Clamp-Crush technique
- Stapler hepatectomy (Experimental)
  Interventions: Procedure: Stapler hepatectomy

INTERVENTIONS:
Procedure: Clamp-Crush technique — The transectional line is marked and the liver capsule is cauterized. The liver parenchyma is then crushed stepwise using a regular Pèan clamp. Vessels and bile ducts are ligated or clipped. Vessels of less than 2mm diameter are coagulated with the irrigated bipolar forceps.
  Arms: Clamp-Crush technique
Procedure: Stapler hepatectomy — The transectional line is marked and the liver capsule is cauterized. For subsequent transection of the hepatic parenchyma, the liver tissue is fractured with a vascular clamp in a stepwise fashion and subsequently divided with endo GIA vascular staplers.
  Arms: Stapler hepatectomy

SUMMARY:
There is clinical uncertainty and ongoing discussion among liver surgeons regarding the optimal method of parenchymal transection in patients undergoing elective hepatic resection. While the clamp-crushing technique still represents the reference technique for routine liver resections, transection of liver parenchyma using vascular staplers may offer a new and safe technique potentially reducing intraoperative blood loss, operation time as well as peri-operative morbidity. As morbidity of patients undergoing hepatic resection remains high, approaches to lower peri-operative complications are urgently required. Due to the lack of evidence it has to be evaluated, if the technique of stapler hepatectomy decreases intraoperative blood loss as a highly relevant predictor of peri-operative complications, patients' hospital stay and finally health care expenditures. These advantages would favor stapler hepatectomy to be applied in routine liver resections. As RCTs are generally considered to generate the most valid scientific evidence on a treatment's effects, the present trial evaluates potential benefits of stapler hepatectomy in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective hepatic resection
* Stapler hepatectomy and clamp-crushing feasible based on preoperative imaging
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Participation in concurrent intervention trials
* Expected lack of compliance
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Weitz, MD, MSc, Principal Investigator — Department of General, Visceral and Transplantation Surgery, University of Heidelberg
Locations (1):
- Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Rahbari NN, Elbers H, Koch M, Vogler P, Striebel F, Bruckner T, Mehrabi A, Schemmer P, Buchler MW, Weitz J. Randomized clinical trial of stapler versus clamp-crushing transection in elective liver resection. Br J Surg. 2014 Feb;101(3):200-7. doi: 10.1002/bjs.9387. Epub 2014 Jan 8. PMID 24402888
- [Derived] Rahbari NN, Elbers H, Koch M, Bruckner T, Vogler P, Striebel F, Schemmer P, Mehrabi A, Buchler MW, Weitz J. Clamp-crushing versus stapler hepatectomy for transection of the parenchyma in elective hepatic resection (CRUNSH)--a randomized controlled trial (NCT01049607). BMC Surg. 2011 Sep 4;11:22. doi: 10.1186/1471-2482-11-22. PMID 21888669